CLINICAL TRIAL: NCT06972511
Title: Apatamide Combined With Maximal Tumor Eradication for Oligometastatic Prostate Cancer, A Prospective Randomized Controlled Trial
Brief Title: Maximal Tumor Eradication for Oligometastatic Prostate Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY2022-022-B
Record Dates: First submitted 2023-04-26; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Oligometastatic Prostate Cancer
MeSH Terms: interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group A (Experimental): neoadjuvant apatamide plus ADT + radical resection of prostate cancer + extended lymph node dissection + radiotherapy of metastases
  Interventions: Combination Product: neoadjuvant apatamide plus ADT + radical resection of prostate cancer + extended lymph node dissection + radiotherapy of metastases
- Control group B (Active Comparator): Standard ADT treatment
  Interventions: Drug: Standard ADT treatment

INTERVENTIONS:
Combination Product: neoadjuvant apatamide plus ADT + radical resection of prostate cancer + extended lymph node dissection + radiotherapy of metastases — neoadjuvant apadamide plus ADT: apadamide 240 mg qd po + leuproprolirelin 3.75mg subcutaneous injection once every month. After 4 months of neoadjuvant therapy, radical prostate cancer + extended lymph node dissection, lymph node dissection to the level of bilateral common iliac arteries, and radiotherapy for metastases was completed within 3 months after surgery.Postoperative adjuvant ADT therapy, regular follow-up until progress to hormone-resistant prostate cancer (CRPC) and then change treatment regimen.
  Arms: Intervention group A
Drug: Standard ADT treatment — leuproprolirelin 3.75mg subcutaneous injection once every month, regular follow-up until progress to hormone-resistant prostate cancer (CRPC) and then change treatment regimen.
  Arms: Control group B

SUMMARY:
In China, the incidence of prostate cancer is increasing in recent years, and it has ranked 5th among common male tumors and 1st in urinary tumors. Unlike developed countries in Europe and the United States, in China, because prostate-specific antigen (PSA) screening has not been widely popularized, and early prostate cancer is mostly asymptomatic, about 13%-26% of prostate cancer patients have progressed to metastatic hormone-sensitive prostate cancer (mHSPC) at the time of initial diagnosis. Compared with localized prostate cancer, the 5-year survival rate of mHSPC is only 29.3%, which is prone to symptoms such as bone pain, pathological fracture, hematuria, and dysuria and seriously decrease the survival and quality of life. As a result, it is of great significance to carry out more refined management of mHSPC, explore more scientific treatment options, and delay the time to CRPC, which is of great significance for improving the prognosis and quality of life of patients and reducing medical burden. However, there is still no standard treatment strategy for OMPC patients which need more clinical exploration.

Treatment of prostate primary in oligometastatic prostate cancer (OMPC) may improve survival and do not significantly increase complications. Radiotherapy showed excellent therapeutic effects on metastatic lesions, prolonged survival and without increasing significant adverse effects. In 2019, The New England Journal of Medicine reported a TITAN study that combining apatamide with ADT for metastatic hormone-sensitive prostate cancer, which significantly reduced the risk of death (82.4% VS 72.5%, P=0.005), and improved progression-free survival (68.2% VS 47.5, P <0.001) without increasing adverse effects of treatment. In 2020, Johns Hopkins University published a phase I clinical study of radical treatment of 12 cases of OMPC. Patients were treated with neoadjuvant docetaxel chemotherapy or abiraterone, combined with radical prostatectomy for primary lesions, and stereotactic radiation for bone metastases to achieve the purpose of complete tumor eradication. Preliminary results showed that no additional complications were found except neutropenic fever in two cases. At the same time, the proportion of PSA maintained undetectable in 1,2,3 years was 12 / 12 (100%), 10 / 12 (83%) and 8 / 12 (67%), respectively, showing good treatment results.

Since 2014, the applicant has rich research experience in the treatment of oligometastatic prostate cancer and our results showed that systemic therapy combined with local tumor reduction therapy can confer a survival benefit for OMPC patients without a significant increase in complications. This clinical trial aimed to analyze the clinical efficacy and safety of maximal tumor eradication strategy for oligometastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 75 years
* EORTC QLQC-30 score 2
* Life expectancy of 10 years
* Patients with oligometastatic prostate cancer on clinicopathological assessment
* Patients are suitable for radiotherapy and prostatectomy surgery
* Patients agree to participate in the study and sign the informed consent form before enrollment

Exclusion Criteria:

* Tumor related fracture
* Cannot accept radiotherapy
* Visceral metastasis
* Serious infection
* Thromboembolism history
* Not effectively controlled cardiovascular complications

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to hormone-resistant prostate cancer （TTCRPC） | 5 years

SECONDARY OUTCOMES:
overall survival rate | 5 years
time to clinical imaging progression in both groups | 5 years
pathological complete response rate | 5 years
minimum PSA after 6 months of treatment in the two groups | 5 years
annual EORTC QLQC-30 score after treatment | 5 years
survival rate of disease-free progression | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- RenJi hospital, school of Medicine, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No